CLINICAL TRIAL: NCT02142777
Title: S-Equol in Alzheimer's Disease (SEAD) Trial
Acronym: SEAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Russell Swerdlow, MD (Other)
Collaborators: Ausio Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor-Investigator, Russell Swerdlow, MD, Gene and Marge Sweeney Professor of Neurology, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00001228
Record Dates: First submitted 2014-05-08; First posted 2014-05-20 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Alzheimer's Disease
Keywords: S-equol; COX activity
MeSH Terms: conditions — Alzheimer Disease | interventions — Equol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Investigational (Experimental): All study subjects will take a 10mg pill by mouth twice daily over a 6 week period. Subjects will receive either placebo or S -Equol. They will not know which they are receiving.
  Interventions: Drug: S -Equol; Drug: Placebo

INTERVENTIONS:
Drug: S -Equol — We will determine if the intervention (S-equol) alters platelet mitochondria COX activity.
  Other Names: AUS-131
Drug: Placebo — The placebo has no active ingredients but is made to look like the study drug.

SUMMARY:
The purpose of this study is to determine if S-equol could benefit persons with Alzheimer's Disease (AD).

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is a progressive brain disorder which causes memory and thinking problems. The exact cause of AD is unknown. Researchers believe mitochondria (the part of your cells that produces energy) might be linked to symptoms of AD. Some studies have shown that patients with Alzheimer's disease have reduced mitochondrial activity or have fewer mitochondria present in neurons. In this study, it is believed that by targeting mitochondria, we might learn more about its influence on AD symptoms.

Mitochondria have a receptor site for estrogen (a hormone) called estrogen receptor β (ERβ). When estrogen attaches to this site, it promotes mitochondrial function. Studies have also suggested ERβ stimulation can cause cells to create new mitochondria. More mitochondria, or increased activity of existing mitochondria, in the cell might have an impact on patients with Alzheimer's disease. One way to measure this increase in function is to look for the presence of an enzyme called COX in your blood. If a drug increases mitochondrial function, there will be an increase in COX concentration in the bloodstream.

By doing this study we hope to learn if S-equol, a compound that acts like estrogen in the body, causes such an increase in mitochondrial activity. We also hope to determine the tolerability of a therapeutic dose of S-equol. It is our goal to advance the understanding of AD, particularly in women.

ELIGIBILITY:
Inclusion Criteria:

* Very mild (CDR 0.5) or mild (CDR 1) AD at time of last KU ADC assessment
* Have a study partner
* Speak English as primary language

Exclusion Criteria:

* No viable study partner
* Report a potentially confounding, serious medical risk such as type 1 diabetes, cancer, or a recent cardiac event (i.e. heart attack, angioplasty, etc.)
* Use any type of estrogen replacement therapy

Ages: 60 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
platelet mitochondria cytochrome oxidase (COX) activity | Change from Baseline to 6 Weeks
  Activity will be identified by the percentage of subjects who show an increase in COX activity while on the active treatment as compared to the COX activity while on placebo.

SECONDARY OUTCOMES:
safety of S-equol | 6 Weeks
  Determine if 10mg twice daily is a safe and well tolerated dose for persons with AD. Safety will be ascertained through the use of a questionnaire that queries a list of standard drug side effects.

CONTACTS AND LOCATIONS:
Overall Officials: Russell H Swerdlow, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States